CLINICAL TRIAL: NCT01304537
Title: Open Label, Proof of Concept, Phase I/II Study of the Safety, Tolerability and Efficacy of Intravenous Alpha-1 Antitrypsin (AAT) [Trade Name Glassia™] in Type 1 Diabetes Mellitus
Brief Title: Study of the Safety and Efficacy of Intravenous Alpha-1 Antitrypsin in Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kamada, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Kamada-AAT (IV) - 008
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2013-02

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — alpha 1-Antitrypsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Alpha-1 Antitrypsin 40mg (AAT, Glassia®) (Experimental): Subjects in this arm will receive a dose of 40 mg/kg throughout the study.
  Interventions: Drug: Alpha-1 Antitrypsin 40mg (AAT, Glassia®)
- Alpha-1 Antitrypsin 60mg (AAT, Glassia®) (Experimental): Subjects in this arm will receive a dose of 60 mg/kg throughout the study.
  Interventions: Drug: Alpha-1 Antitrypsin 60mg (AAT, Glassia®)
- Alpha-1 Antitrypsin 80mg (AAT, Glassia®) (Experimental): Subjects in this arm will receive a dose of 80 mg/kg throughout the study.
  Interventions: Drug: Alpha-1 Antitrypsin 80mg (AAT, Glassia®)

INTERVENTIONS:
Drug: Alpha-1 Antitrypsin 40mg (AAT, Glassia®) — Each study group will undergo 3 treatment periods:12 weeks, 8 weeks and 4 weeks.
  Arms: Alpha-1 Antitrypsin 40mg (AAT, Glassia®)
Drug: Alpha-1 Antitrypsin 60mg (AAT, Glassia®) — Each study group will undergo 3 treatment periods:12 weeks, 8 weeks and 4 weeks.
  Arms: Alpha-1 Antitrypsin 60mg (AAT, Glassia®)
Drug: Alpha-1 Antitrypsin 80mg (AAT, Glassia®) — Each study group will undergo 3 treatment periods:12 weeks, 8 weeks and 4 weeks.
  Arms: Alpha-1 Antitrypsin 80mg (AAT, Glassia®)

SUMMARY:
Alpha-1 Antitrypsin (AAT), trade name (Glassia ®), is being explored in this phase I/II trial as a potential disease modifying agent in Type 1 Diabetes Mellitus (T1DM) based on its anti-inflammatory properties. AAT is an acute stress reactant protein that increases during inflammation. In T1DM inflammation serves a major role in disease progression.

DETAILED DESCRIPTION:
AAT is a protein produced by the human liver and secreted into the blood circulation. AAT, which belongs to a group of serine protease inhibitors (SERPINS) is an acute stress reactant protein that increases during stress conditions, including inflammation. AAT blocks serine proteases that enhance pro-inflammatory mediators (i.e. IL-1 alpha, IL-6, IL-8, TNFalpha) as well as induces production of anti-inflammatory mediators (i.e. IL-10 and IL-1-receptor antagonist).

In Type 1 Diabetes Mellitus (T1DM) inflammation serves a major role in disease progression. The inflammatory signature pattern in these patients appears to have been present years before clinical onset.

Although circulating levels of AAT in T1DM are normal, in majority of cases, the activity of AAT is severely compromised by non-enzymatic glycations, supporting the conclusion that serum protease inhibitory capacity is reduced in T1DM.

It has been shown in different studies, including in vivo and in vitro that AAT has a protective affect on pancreatic islets. This has been demonstrated in both decrease in progression of diabetes in the non-obese diabetic (NOD) mouse as well as during transplantation of islets which presented viability and activity (insulin production) in the presence of AAT. More specifically, islet cells are protected by human AAT from apoptosis, as shown by reduced caspase-3 activity after the addition of human AAT to islet culture media.

Based on the mentioned anti-inflammatory properties of AAT sided to in vivo and in vitro studied indicating that AAT may serve as a disease modifying agent in T1DM, the presented study is suggested.

ELIGIBILITY:
Inclusion Criteria:

* Subject (or parent/guardian) willing and able to sign an informed consent
* Age 10-25 (inclusive) years
* Diagnosed with T1DM within the previous 6 months
* Level of C-peptide ≥ 0.2 pmol/mL during MMTT(maximal level)
* Positive for at least one diabetes-related autoantibody(except for insulin autoantibody)
* No significant abnormalities in serum hematology,serum chemistry according to the Investigator's judgment, taking into considerations the potential effects of the diabetic illness.
* No significant abnormalities in urinalysis according to the Principal Investigator's judgment, taking into considerations the potential effects of the diabetic illness.
* No significant abnormalities in ECG per investigator judgment
* Negative for HBsAg and antibodies to HCV, HIV-1
* Non-pregnant, non-lactating female patients, whose screening pregnancy test is negative and who are using contraceptive methods deemed reliable by the investigator.

Exclusion Criteria:

* Subjects who have received an active/ live virus vaccine within 4 weeks of the screening date
* Subjects who have received treatment with corticosteroid medication within 2 months prior to screening or any immunosuppressant or cytostatic agent within 6 months prior to screening
* IgA deficient subjects
* Individuals with a history of severe immediate hypersensitivity reactions, including anaphylaxis, to plasma products
* Planned major surgery within the study period
* Clinically significant intercurrent illnesses, including(but not limited to): cardiac, hepatic, renal,neurological, hematological, neoplastic, immunological, skeletal or other) that in the opinion of the investigator, could interfere with the safety, compliance or other aspects of this study. Patients with well-controlled, chronic diseases could be possibly included after consultation with the treating physician and the sponsor.
* Pregnant or lactating women at entry to study and those who are unwilling to agree to continue to use acceptable methods of contraception throughout the study.
* Presence of psychiatric/ mental disorder or any other medical disorder which might impair the patient's ability to give informed consent or to comply with the requirements of the study protocol.
* Evidence of ongoing viral infection with HCV, HBV and/or HIV-1.
* Evidence of alcohol abuse or history of alcohol abuse or illegal and/or legally prescribed drugs.
* Participation in another interventional clinical trial within 30 days prior to baseline visit.
* Inability to attend scheduled clinic visits and/or comply with the study protocol.
* Any other factor that, in the opinion of the investigator, would prevent the patient form complying with the requirements of the protocol.
* Current use of any medication known to influence glucose tolerance (e.g., beta-blockers, angiotensin-converting enzyme inhibitors, interferons, quinidine anti-malarial drugs, lithium, niacin).
* Current or prior (within the last 30 days prior to screening visit) use of metformin, sulfonylureas, glinides, thiazolidinediones, exenatide, liraglutide, DPP-IV inhibitors or amylin.

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2011-06; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | Approximately 1 year
  Safety and Tolerability: assessed by vital signs(systolic/diastolic blood pressure and heart rate), physical examination, routine safety lab tests, AEs and SAEs.

SECONDARY OUTCOMES:
Efficacy | Approximately 1 year
  Pancreatic beta cell function ; External Insulin dose requirements; Glycosylated hemoglobin (HbA1c) levels.

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Rachmiel, B.Med.Sc, Principal Investigator — Assaf Haroffeh Medical Center, Zerifin, Israel; Yael Lebenthal, MD, Principal Investigator — Institute for Endocrinology & Diabetes, Schneider Children's Medical Center, Israel
Locations (2):
- Israel (2):
  - Institute for Endocrinology and Diabetes, National Center for Childhood Diabetes at Schneider Children's Medical Center of Israel, Petah Tikva, Israel
  - Assaf Haroffeh Medical Center, Ẕerifin, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ozeri E, Mizrahi M, Shahaf G, Lewis EC. alpha-1 antitrypsin promotes semimature, IL-10-producing and readily migrating tolerogenic dendritic cells. J Immunol. 2012 Jul 1;189(1):146-53. doi: 10.4049/jimmunol.1101340. Epub 2012 May 25. PMID 22634621